CLINICAL TRIAL: NCT04755348
Title: A Single Dose, Randomised, Crossover Study to Assess the Pharmacokinetics of Oral Nicotine Pouches and Lozenges in Healthy Adults
Brief Title: A Study to Assess the Pharmacokinetics of Oral Nicotine Pouches and Lozenges in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British American Tobacco (Investments) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BAT2221030
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Tobacco Use; Tobacco Smoking; Cigarette Smoking
MeSH Terms: conditions — Tobacco Use; Tobacco Smoking; Cigarette Smoking | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Product usage order ABFCED (Experimental): Subjects will use each of the 6 products (ABFCED) during an familiarization period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F
- Product usage order BCADFE (Experimental): Subjects will use each of the 6 products (ABECD) during an familiarization period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F
- Product usage order CDBEAF (Experimental): Subjects will use each of the 6 products (CDBEAF) during an familiarization period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F
- Product usage order DECFBA (Experimental): Subjects will use each of the 6 products (DECFBA) during an familiarization period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F
- Product usage order EFDACB (Experimental): Subjects will use each of the 6 products (EFDACB) during an familiarization period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F
- Product usage order FAEBDC (Experimental): Subjects will use each of the 6 products (FAEBDC) during an familiarization period, followed by a 4 hour Test Session
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D; Other: Product E; Other: Product F

INTERVENTIONS:
Other: Product A — A 4mg nicotine pouch product
Other: Product B — A 4mg nicotine pouch product
Other: Product C — A 2mg nicotine lozenge product
Other: Product D — A 2mg nicotine lozenge product
Other: Product E — A 2mg nicotine lozenge product
Other: Product F — A 2mg nicotine lozenge product

SUMMARY:
This is a randomised, open-label, confined, cross-over study to evaluate the nicotine pharmacokinetics (PK) of modern oral nicotine pouches and nicotine lozenges carried out in 36 healthy adult subjects who smoke cigarettes and who may have experience using smokeless tobacco (loose or pouches).

DETAILED DESCRIPTION:
Starting on Day 1, subjects will check-in at the clinical site to complete procedures to confirm eligibility. Following basic check-in procedures (e.g., urine pregnancy test, urine drug screen, alcohol test and vital signs), subjects will continue with a 7-day confinement. Subjects will be randomized to a product sequence (using a Williams design).

Test sessions will occur every day during the remainder of the study. The active period of each test session will last for approximately 4 hours after the start of Investigational Product (IP) use. During each test session, a subject will be required to use their randomized IP and during the session, PK blood draws and a subjective effects questionnaire will be collected.

The day prior to each test session, subjects will participate in a product familiarization period in which they will use one pouch or lozenge of their randomized IP. The product familiarization period will occur after the scheduled test session (or after enrollment and randomization on Day 1) and before the 12-hour tobacco and nicotine abstinence period. Subjects should use the IP pouch for at least 30 minutes or allow the lozenge to dissolve slowly.

Subjects will provide usual brand (UB) cigarettes for use during study confinement and have access to their UB cigarettes for ad libitum use with the exception of 1) during the test session, 2) during the the minimum 12-hour tobacco and nicotine abstinence period prior to each test session and 3) a minimum of one hour after IP use during the product familiarization period. Each UB cigarette must be requested from site staff and used butts returned to site staff for accountability.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy males or females, 21 to 60 years of age, inclusive, at the time of consent.
3. Smoke manufactured combustible, filtered, non-menthol or menthol cigarettes, 83 mm to 100 mm in length as primary source of tobacco.
4. Smokers who self-report use of a smokeless tobacco product (loose or pouch) prior to screening may also be enrolled.
5. Smokes an average of at least 10 cigarettes per day (CPD) and inhale the smoke, for at least 6 months prior to screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of screening), or clinical study participation (prior to 30 days of screening) will be allowed at the discretion of an investigator.
6. Agrees to smoke the same Usual Brand (UB) cigarette throughout the study period. The UB cigarette is defined as the reported cigarette brand and style currently smoked most frequently by the subject. If a subject reports use of a different UB cigarette at check in, that subject may continue provided they use that same UB cigarette throughout the study.
7. Expired breath carbon monoxide (ECO) level is ≥ 10 ppm and ≤ 100 ppm at screening.
8. Positive urine cotinine test at screening.
9. Willing to use the UB cigarette and nicotine pouch or lozenge IPs during the study period.
10. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to start of each of six test sessions.
11. If female and of non-childbearing potential, must meet one of the following criteria:

    1. Surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation/occlusion); or
    2. In a menopausal state (at least 1 year without menses), as confirmed by follicle stimulating hormone (FSH) levels (≥40 mIU/mL).
12. If female and of childbearing potential, must agree to use one of the accepted contraceptive regimens from at least 30 days prior to the first administration of the IP during the study, and for at least 30 days after the last dose of the IP. An acceptable method of contraception includes one of the following:

    1. Abstinence from heterosexual intercourse;
    2. Hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch);
    3. Intrauterine device (with or without hormones); or
    4. Use of a double barrier method (e.g., condom and spermicide) during the study and for at least 30 days after the last dose of the study medication.
13. Agrees to an in-clinic confinement of 7 days (6 nights).

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of an investigator, makes the study subject unsuitable to participate in this clinical study.
2. History, presence of, or clinical laboratory test results indicating diabetes.
3. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the screening visit. As-needed treatment, such as inhalers, may be included at an investigator's discretion pending approval from the Medical Monitor.
4. History or presence of bleeding or clotting disorders.
5. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
6. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes at screening and at check-in Day 1.
7. Weight of ≤ 110 pounds.
8. Hemoglobin level is < 12.5 g/dL for females or <13.0 g/dL for males at screening.
9. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
10. Positive urine drug screen without evidence of a prescription or urine alcohol test at Day 1 (check-in), with the exception of for tetrahydrocannabinol (THC). If positive for THC, a cannabis intoxication evaluation will be performed at check-in, and inclusion will be at the discretion of an investigator.
11. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
12. Self reports use of the study IP (nicotine pouches or lozenges) currently or in the past.
13. Recreationally uses vapor products (e.g., e-cigarettes, tank systems) more than one day per week, for the past 6 months prior to screening.
14. Current, regular user (i.e., > 5 times per month) of any tobacco products other than combustible cigarettes or smokeless tobacco within the last 6 months prior to screening.
15. Use of any medication or substance that aids in smoking cessation, including but not limited to any nicotine replacement therapy (NRT) (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
16. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or self-reports a previous attempt within (≤) 30 days prior to the signing the informed consent.
17. Any use of aspirin (≥ 325 mg/day) or anticoagulants within (≤) 30 days prior to the signing of informed consent.
18. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
19. Whole blood donation within 8 weeks (≤ 56 days) prior to the signing of informed consent and between screening and check-in Day 1.
20. Plasma donation within (≤) 7 days prior to the signing of informed consent and between screening and check-in Day 1.
21. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
22. Participation in another clinical trial within (≤) 30 days prior to the signing of informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing of informed consent in the current study.
23. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol result at screening or check-in Day 1.
24. Determined by an investigator to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Cmax | 240 minutes
  Maximum baseline-adjusted plasma concentration of nicotine
AUC0-240 mins | 0-240 minutes
  Baseline-adjusted area under the plasma nicotine concentration-versus-time curve from time zero to 240 minutes after the start of IP use

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Altasciences Clinical Kansas, Inc.
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No